CLINICAL TRIAL: NCT07115212
Title: Effectiveness of Bromelain Supplement in Reduction of Facial Swelling Caused by Orthognathic Surgery
Brief Title: Bromelain for Post-surgery Facial Swelling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Bazina (Other)
Responsible Party: Sponsor-Investigator, Mohamed Bazina, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 99500
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Malocclusion
Keywords: Bromelain; Oral Supplements
MeSH Terms: conditions — Malocclusion | interventions — Bromelains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bromelain Supplement (Experimental): 1000mg bromelain supplement once a day, 2 days prior to and 7 days following surgery
  Interventions: Dietary Supplement: Bromelain
- Control (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Bromelain — 1 tablet daily with water, for 9 days-starting 2 days before surgery and continuing for 7 days after. Record each dose in the provided log, along with any other medications taken and the time they were taken.
  Other Names: Naturebell
  Arms: Bromelain Supplement

SUMMARY:
The goal of this clinical trial is to learn if Bromelain Supplement works to decrease the amount of swelling or the amount of time swelling is present following jaw surgery. It will also learn about the safety of Bromelain supplement. The main questions it aims to answer are:

Does Bromelain decrease facial swelling following orthognathic, or jaw, surgery? Does Bromelain supplement decrease the amount of time that patients are swollen following orthognathic, or jaw, surgery?

Participants will:

Take Bromelain supplement once daily for 9 days total. Take 2 days before surgery and 7 days following surgery.

Keep a log of when the bromelain supplement is taken as well as another other medications.

Visit the clinic with pre and post surgical protocol

ELIGIBILITY:
Inclusion Criteria:

* undergoing orthognathic surgery

Exclusion Criteria:

* craniofacial anomalies
* incomplete patient data
* systemic disease that could affect healing
* allergy to latex or pineapple
* under 18 years of age
* non english speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Volume of Swelling | Baseline, and post intervention weeks 1, 2, 4, and months 3 and 6
  Images will be obtained with the Vectra 3D imaging system to look at the volume of swelling in patients that undergo orthognathic surgery and measured in Cubic Centimeters. Will also have a heat map to visually show where swelling has increased or decreased since previously obtained imaging. All these images and measurements will be compared between the control and experimental groups.
Duration of Swelling following Orthognathic Surgery | Baseline, and post intervention weeks 1, 2, 4, and months 3 and 6
  Images will be obtained with the Vectra 3D imaging system to look at the volume of swelling in patients that underwent orthognathic surgery at multiple time periods. With comparisons of these multiple photos the duration of swelling can be assessed and compared to the average amount of time it takes swelling to go down in a patient not taking bromelain supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bazina, DDS, MSD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No